CLINICAL TRIAL: NCT01627678
Title: Immunotherapy of HIV-infected Patients An Open, Dose-escalating Assessment of Vacc-C5 With Either GM-CSF or Alhydrogel as Adjuvant in HIV-1-infected Subjects on Antiretroviral Therapy (ART)
Brief Title: Immunotherapy With Vacc-C5 With Adjuvant GM-CSF or Alhydrogel in HIV-1-infected Subjects on ART
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bionor Immuno AS (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTN-BI-Vacc-C5-2011/1; 2012-000710-11 (EudraCT Number)
Record Dates: First submitted 2012-06-21; First posted 2012-06-26 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: HIV-1 Infection
Keywords: HIV-1, Vacc-C5
MeSH Terms: interventions — sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1= Arm A: Vacc-C5 /GM-CSF. (Experimental): Arm 1=Arm A: Vacc-C5 with GM-CSF as adjuvant administered intradermally.
  Interventions: Drug: Vacc-C5/GM-CSF
- Arm 2=Arm B: Vacc-C5/Alhydrogel (Experimental): Arm 2=Arm B: Vacc-C5 with Alhydrogel as adjuvant administered intramuscularly.
  Interventions: Drug: Vacc-C5/Alhydrogel

INTERVENTIONS:
Drug: Vacc-C5/GM-CSF — Arm 1=Arm A: Vacc-C5 with GM-CSF as adjuvant administered intradermally.
  Other Names: Vacc-C5 = C5-peptide; GM-CSF = Leukine
  Arms: Arm 1= Arm A: Vacc-C5 /GM-CSF.
Drug: Vacc-C5/Alhydrogel — Arm 2=Arm B: Vacc-C5 with Alhydrogel as adjuvant administered intramuscularly.
  Other Names: Vacc-C5 = C5-pepide; Alhydrogel = Aluminum-containing adjuvant
  Arms: Arm 2=Arm B: Vacc-C5/Alhydrogel

SUMMARY:
Background:

Despite the introduction of highly effective antiretroviral therapy (ART) regimes, which control the HIV infection and results in increases in CD4 cell counts and an undetectable viral load, many patients suffer from increased morbidity. There is evidence that presence of antibodies against the C5 region of gp120 strongly correlates with slower disease progression, and that loss of antibody responses to this region are associated with progression.

Investigational product:

Vacc-C5 is a single heterodimeric peptide-based HIV therapeutic vaccine corresponding to the C5 region on gp120 and the external domain of gp41. The vaccine is intended to create a non-neutralizing antibody against C5 region.

Study objectives:

1. To evaluate safety of the vaccination regimens
2. To evaluate C5-specific humoral immune responses (antibodies), T cell responses, T cell activation markers and other immune markers.

DETAILED DESCRIPTION:
Background:

Despite the introduction of highly effective antiretroviral therapy (ART) regimes, which control the HIV infection and results in increases in CD4 cell counts and an undetectable viral load, many patients suffer from increased morbidity. There is evidence that presence of antibodies against the C5 region of gp120 strongly correlates with slower disease progression, and that loss of antibody responses to this region are associated with progression.

Investigational product:

Vacc-C5 is a single heterodimeric peptide-based HIV therapeutic vaccine corresponding to the C5 region on gp120 and the external domain of gp41. The rationale behind the Vacc-C5 is the finding that long-term non-progressors (LTNP) subjects have more antibodies towards the C5 part of gp120 than HIV infected subjects with a more rapid disease progression.

The primary objective of Vacc-C5 immunotherapy is to induce a humoral immune response. The vaccine is intended to create a non-neutralizing antibody against the C5 region and to thereby mimic a natural process in HIV-infected long-term non-progressors (LTNP) subjects.

Use of adjuvant:

Peptide vaccines are poorly immunogenic by themselves. To induce measurable levels of T helper cell type 1 (Th1) or type 2 (Th2) immune responses against these peptides, an adjuvant is often required.

Two different adjuvants are to be used in this study:

1. GM-CSF which facilitates dendritic cell maturation and migration to the lymph nodes for antigen presentation. The regimen when using this adjuvant is intradermal administration.
2. Aluminum-containing adjuvants is well known. They have been administered to human beings and animals in millions of doses of vaccines. This type of vaccine is usually administered intramuscularly or subcutaneously. In this study intramuscular administration will be used.

Primary objective:

It is to evaluate the safety of Vacc-C5 at three different dose levels given intradermally with GM-CSF as adjuvant or given intramuscularly with Alhydrogel as adjuvant.

Secondary objectives:

1. To evaluate C5-specific humoral immune responses (antibodies).
2. To evaluate the C5-specific T cell responses by ELISPOT and T cell proliferation.
3. To evaluate T cell activation markers (e.g. CD38, HLA-DR) and other immune markers.

Study design:

The study is an open, dose-escalating, single centre study in HIV-positive subjects on treatment (ART). Two different vaccine regimens will be tested:

1. Arm A: Vacc-C5 with GM-CSF as adjuvant administered intradermally.
2. Arm B: Vacc-C5 with Alhydrogel as adjuvant administered intramuscularly.

Three dose levels of Vacc-C5 (100, 300 and 900 microgram will be tested for each of the two vaccination regimen. A dose escalation design (3+3) will be used, and if no dose limiting toxicity (DLT) is detected 18 subjects will be included in each arm.

Subjects who have been HIV-positive and stable on ART for the last 6 months with CD4 cell counts ≥400x 10 6 /L and who meet the other inclusion and exclusion criteria will be eligible for the study. The duration of the study is 26 weeks plus a screening period of up to 12 weeks.

During the Treatment Period, all subjects will remain on their ART and receive three immunizations; at Weeks 1, 2 and 4, with Vacc C5 including either GM-CSF or Alhydrogel as adjuvant.

The study is sequential, meaning that the first three subjects in each arm receive the lowest dose (three subjects) 100 µg Vacc-C5. If no dose limiting toxicity has been detected after week 4 vaccination, three more subjects will be added and the next dose level will be started.

ELIGIBILITY:
Inclusion Criteria:

* Age between18 years and 55 years, both genders.
* HIV positive at least one year.
* Clinically stable on ART for the last 6 months (changes in therapy is allowed as long as the viral load is stable).
* Documented viral load (HIV-1 RNA) less than 50 copies/mL for the last six months. Single blips (up to 500 copies/mL) are allowed.
* Documented pre-study CD4 cell count ≥ 400x106/L for at least six months (if below at screening, a re-analysis is allowed).
* Nadir (lowest ever) CD4 cell count ≥ 200x106/L (nadir below 200x106/L requires two consecutive analyses).
* Signed informed consent.

Exclusion Criteria:

* Reported pre-study AIDS-defining illness within the previous year
* Malignant disease.
* On chronic treatment with immunosuppressive therapy.
* Unacceptable values of the hematologic and clinical chemistry parameters, as judged by the Principle Investigator (or designee), including creatinine values >1.5x upper limit of normal (ULN), and AST (SGOT), ALT (SGPT) and alkaline phosphatase values >2.5x ULN.
* Concurrent chronic active infection such as viral hepatitis B or C or tuberculosis.
* Pregnant or breastfeeding women.
* Women of childbearing potential not using reliable and adequate contraceptive methods (defined as: use of oral, implanted, injectable, mechanical or barrier products for the prevention of pregnancy; practicing abstinence; sterile) during the study, or sexually active male subjects with partners of childbearing potential unwilling to practice effective contraception during the study.
* Current participation in other clinical therapeutic studies.
* Incapability of compliance to the treatment protocol, in the opinion of the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Safety measured as change of AE records, clinical chemistry (incl. CD4, CD8, HIV-1 RNA)and hematology laboratory elevations | From screening and week 1 to weeks 2, 4, 6, 12, 13, 15, 21, 22 and 26
  * AEs recorded at each scheduled and unscheduled visit.
  * Concomitant medications recorded at each scheduled visit.
  * Vital signs (heart rate, blood pressure) at screening, weeks 1, 4, 6, 12, 13, 15, 21, 22 and 26 (End of study).
  * Weight at screening and weight at weeks 1, 12 and 26 (End of study).
  * Clinical laboratory evaluations (clinical chemistry, hematology) at screening, weeks 1, 4, 6, 12, 15, 21 and 26 (End of study).
  * Viral load (HIV-1 RNA) at screening, weeks 1, 6, 15 and 26 (End of study).
  * Urine stix at weeks 1, 4, 6, 12, 15, 21 and 26 (End of study).

SECONDARY OUTCOMES:
Change in Humoral and T cell responses | From screening and week 1 to weeks 4, 6, 12, 13, 15, 21, 22 and 26
  * Humoral immune response - C5 antibody level at screening, weeks 1, 4, 6, 12, 13, 15, 21, 22 and 26 (End of study).
  * B cell antibody level at weeks 1, 6, 13 and 22.
  * T cell response and activation markers (e.g. CD38, HLA-DR) and other immune markers at weeks 1, 6, 15and 26 (End of study).

CONTACTS AND LOCATIONS:
Overall Officials: Vidar Wendel-Hansen, MD PhD, Study Director — Bionor Pharma AS
Locations (1):
- Oslo University Hospital, Ullevål, Oslo, Norway

REFERENCES:
- [Derived] Brekke K, Sommerfelt M, Okvist M, Dyrhol-Riise AM, Kvale D. The therapeutic HIV Env C5/gp41 vaccine candidate Vacc-C5 induces specific T cell regulation in a phase I/II clinical study. BMC Infect Dis. 2017 Mar 24;17(1):228. doi: 10.1186/s12879-017-2316-x. PMID 28340570